CLINICAL TRIAL: NCT04855903
Title: Rehabilitation of Executive Functions in the Activities of the Daily Living of Chronic Post-stroke Patients: Using Virtual Reality and Computerized Rehabilitation to Simulate Real Environment for Rehabilitation.
Brief Title: Executive Functions Computerized Rehabilitation Using Virtual Reality to Improve Activities of Daily Living Post-stroke
Acronym: RéFEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC31/19/0552
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: N-of-1 trials; cognitive rehabilitation; computerized rehabilitation; virtual reality; executive functions; occupational therapy; post-stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Multiple Baseline case experimental design (N-of-1 trial)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (early phase B) (Experimental): 2 phases of cognitive training: Phase A : rehabilitation program in standard ergotherapy during 3 weeks Phase B : cognitive training using Covirtua Cognition software during 4 weeks
  These 2 phases will be followed by a follow-up phase during 5 weeks
  Interventions: Device: Covirtua Cognition software
- Arm 2 (mid phase B) (Experimental): 2 phases of cognitive training: Phase A : rehabilitation program in standard ergotherapy during 4 weeks Phase B : cognitive training using Covirtua Cognition software during 4 weeks
  These 2 phases will be followed by a follow-up phase during 4 weeks
  Interventions: Device: Covirtua Cognition software
- Arm 3 (late phase B) (Experimental): 2 phases of cognitive training: Phase A : rehabilitation program in standard ergotherapy during 5 weeks Phase B : cognitive training using Covirtua Cognition software during 4 weeks
  These 2 phases will be followed by a follow-up phase during 3 weeks
  Interventions: Device: Covirtua Cognition software

INTERVENTIONS:
Device: Covirtua Cognition software — Cognitive training with Covirtua Cognition software

SUMMARY:
This research aims to evaluate the effects of a cognitive reeducation carried out with the COVIRTUA Cognition software using a virtual environment, on real-life execution of activities of daily living (ADL) for patients with post-stroke dysexecutive disorders. We will assess patients' performances in achieving ADLs by the Goal Attainment Scaling (GAS) throughout the follow-up (3 months), based on the goals set at the beginning of management with each patient.

DETAILED DESCRIPTION:
Many post-stroke patients, especially those with frontal lobe lesions, have chronic impairments in mental flexibility, leading to difficulties in decision-making, action planning, or behavioural perseverance. Techniques for remediation of these dysexecutive disorders are often performed in a hospital or in a liberal office. The possible progress resulting from this rehabilitation is rarely transposed into the patient daily life performances, executed in a richer and less controlled environment than the usual place of re-educational. Here, we wish to assess the effective benefits (i.e. in carrying out the activities of daily living) of a computerized rehabilitation program addressing executive functions and based on virtual reality, simulating ADLs. We use in this study a multiple baseline single case experimental design (AB design with a follow-up beyond), including for each patient: pretreatment (phase A), treatment (phase B), and follow-up phase.

Pretreatment includes a routine sensitivomotor neurological rehabilitation program that doesn't specifically target executive functions in daily living activities (3 to 5 weeks depending on randomization). Treatment consists in a 4 weeks virtual reality cognitive training program, including four 45-minute sessions per week with an occupational therapist for cognitive rehabilitation in a virtual environment with the COVIRTUA Cognition software. The follow-up phase (5 to 3 weeks depending on randomization) includes no support for executive functions, either in a rehabilitation centre or in a liberal office.

ELIGIBILITY:
Inclusion Criteria:

* Vascular brain injury (stroke), in chronic phase (6 months or more after stroke), responsible for dysexecutive syndrome authenticated by the GREFEX/GRECO battery (Executive Function Evaluation Reflection Group)
* Men and women over the age of 18
* Presence of a caregiver
* Social Security affiliation
* Signing free and informed consent following clear and detailed information
* Sufficient understanding of the French language to participate in the study

Exclusion Criteria:

* Pregnant women (clinical examination)
* Alcohol and/or narcotics addiction
* Major hearing deficit
* Major visual deficit
* Neurological pathology other than stroke or psychiatric disorder
* Unstable epilepsy
* Patient undergoing rehabilitation at a liberal therapist targeting executive functions during study time
* Patient under safeguard of justice.
* Patient simultaneously participating in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Evolution of performance at GAS (Goal Attainment Scaling) | T3 months
  Performance in carrying out activities of daily living will be evaluated in an ecological situation using Kiresuk and Sherman's 'Goal Attainment Scaling' (GAS) method. The individual goals to be achieved and performance levels of the GAS will be determined at inclusion, and evaluated twice a week during the three phases (A, B and follow-up phase). The primary outcome will be the evolution of the GAS score evaluated twice a week during 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CATELLA, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - Centre de la Tour de Gassies, Bruges
  - Hôpital Swynghedauw, Lille
  - University hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No